CLINICAL TRIAL: NCT05780827
Title: Analysis of Clinical Data of Patients With Temporomandibular Joint Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Meiqing Wang, Professor, State Key Laboratory of Military Stomatology, Department of Oral Anatomy and Physiology, School of Stomatology, Air Force Military Medical University, China
Other Study IDs: Oral Anatomy & Physiology AFMU
Record Dates: First submitted 2023-02-16; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Postural Balance; Occlusion
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: No symptoms and signs of oral and maxillofacial dysfunction are required
- Patients with temporomandibular joint disorder: Patients with temporomandibular joint disorder

SUMMARY:
According to our previous research and clinical observation results, the motor function of the oral, maxillofacial and cervical body is closely related to the occlusal contact. Not only that, the occlusal contact also affects the psychological activities related to movement. There are many technical means to evaluate the occlusion clinically. However, the occlusion is a complex motor organ with more than 3 dimensional (including age factors) morphological characteristics, which makes the occlusion have obvious individualized characteristics. It is of great significance to objectively evaluate oral health to accurately extract occlusal contact features, analyze the relationship between occlusion and the motor function of oral, maxillofacial, neck and body as well as the corresponding psychological characteristics, and establish an evaluation method of occlusal function for evaluating motor function and psychological characteristics.

DETAILED DESCRIPTION:
The project is intended to carry out the correlation between occlusal contact and subclinical indicators of physical and mental health. The data collection method combining occlusal detection, physical fitness detection and questionnaire survey is adopted to obtain the target data, and then the machine learning method is used to extract the sensitive technical parameters from the collected data.

1. Data collection

1. 3D occlusal contact detection: It is planned to recruit 1000 healthy volunteers and use "oral laser scanner" to conduct 3D scanning on them, so as to obtain 3D occlusal digital model data of 1000 healthy volunteers. A control group was set up at the same time, and the model and data of 10000 patients who had previously visited the hospital in our department's existing case database were used for comparative analysis.
2. Physical fitness test: for the dynamic/static standing balance function test of volunteers, the dynamic/static balance test system developed by our research group is used to test and obtain physical fitness parameters. The sample size is statistically estimated, and the average number of dynamic/static tests is not less than 50. A control group was established at the same time: volunteers with temporomandibular joint disorder and abnormal occlusion.
3. Psychological evaluation: including volunteers' personality characteristics, mental health level and basic flight ability.

2. The extraction of machine learning occlusal parameters uses the 3D occlusal evaluation system reported by us to calculate the occlusal tightness, and extracts the three-dimensional direction and comprehensive parameters of the upper and lower jaw according to the method reported by us, a total of 10 quantitative indicators.

3. Correlation analysis of occlusal contact and physical and mental health indicators For the collected occlusal parameter data, the physical parameter data obtained from the dynamic/static orthostatic balance function test, and the psychological parameter data obtained from the personality characteristics, mental health level and other tests, the difference of the dynamic/static ability of volunteers with healthy, temporomandibular joint disorder and abnormal occlusion was compared with the analysis of variance; Multiple regression method was used for correlation test; Machine learning is used for cluster analysis.

ELIGIBILITY:
Experimental group

Inclusion Criteria:

No symptoms and signs of oral and maxillofacial dysfunction.

Exclusion Criteria:

1. Those who have received orthodontic treatment
2. Have a history of maxillofacial trauma
3. Maternity
4. Those who take any medicine for a long time
5. Patients with chronic diseases such as tumors, endocrine diseases, psychosocial diseases and immune diseases.
6. Other persons who are unable to cooperate with the project by themselves, such as action barriers.

Control group

Inclusion Criteria:

Suffer from symptoms and signs of oral and maxillofacial dysfunction

Exclusion Criteria:

1. Those who have received orthodontics or other treatment
2. Have a history of maxillofacial trauma
3. Maternity
4. Those who take any medicine for a long time
5. Patients with chronic diseases such as tumors, endocrine diseases, psychosocial diseases and immune diseases.
6. Other persons who are unable to cooperate with the project by themselves, such as action barriers.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Advertisements were issued in universities and stomatological hospitals to recruit healthy volunteers and patients with temporomandibular joint.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Postural Balance | 2023.02.16-2023.12.31
  Use the "balance tester" to measure the dynamic and static measurement data of "healthy volunteers" and "patients with TMD", and carry out the homogeneity test of variance for the obtained measurement data. If it is subject to the homogeneity of variance, carry out the group t-test or analysis of variance for the data, and compare the differences between groups and within groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wang MeiQing, M.D, Study Director — Professor, State Key Laboratory of Military Stomatology, Department of Oral Anatomy and Physiology, School of Stomatology
Locations (1):
- Forth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No